CLINICAL TRIAL: NCT02851758
Title: Transplantation of Autologously Derived Mitochondria for Protection Against Ischemia-reperfusion Injury Following Ischemia in Subjects on ECMO Support
Brief Title: Transplantation of Autologously Derived Mitochondria Following Ischemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sitaram Emani, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00014558
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Extracorporeal Membrane Oxygenation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous mitochondria injection (Experimental): All subjects will have autologous mitochondria injected into ischemic areas of the myocardium (via injection or infusion).
  Interventions: Other: autologous mitochondria transplantation

INTERVENTIONS:
Other: autologous mitochondria transplantation — Autologous mitochondria obtained from the subject's own skeletal muscle will be injected or infused into the ischemic myocardium

SUMMARY:
The investigators propose a robust therapeutic intervention to ameliorate myocardial ischemia/ reperfusion injury and significantly decrease morbidity and mortality in patients requiring extracorporeal membrane oxygenation (ECMO), by direct injection of autogeneic mitochondria into the ischemic myocardium.

DETAILED DESCRIPTION:
Autologous mitochondria will be delivered to the ischemic heart muscle in one of two ways, during clinically indicated surgical procedure or during clinically indicated cardiac catheterization.

For surgical re-operation subjects:

After the subject's chest is open, 1-2 6mm biopsies will be collected from the exposed skeletal muscle of the chest wall. The tissue will be processed at bedside to extract the autologous mitochondria. Surgery will proceed as clinically indicated. Prior to closure of the chest, autologous mitochondria will be injected via 5-10 injections of approximately 0.1 mL each to the damaged area (if damaged muscle is local) or via injection into the proximal aorta while cross-clamped for clinically indicated surgery for global distribution of mitochondria via the coronary arteries if there is no evident area of damage. Following completion of surgical maneuvers the mitochondria will be injected into the aorta and the cross-clamp will be removed. If there is global injury but a cross-clamp is not clinically indicated, direct injection into the myocardium will occur throughout the ventricle as previously described. Chest closure will then occur as and if clinically indicated for both techniques.

For catheterization subjects:

Once in the catheterization lab, the temporary chest closure will be removed and 1-2 6 mm biopsies will be collected from the exposed skeletal muscle of the chest wall by the cardiac surgery team. The tissue will be processed at bedside to extract the autologous mitochondria. The catheterization will proceed as clinically indicated. Prior to completion of the procedure (interventional to restore blood flow or hemodynamics), mitochondria will be infused in 5 mL of buffer as conducted in large animal studies (5) via intracoronary infusion followed by a 5 mL flush with normal saline. Total dose of mitochondria will be equal to direct injection subjects, with a larger dilution to allow to infusion via cardiac catheter.

If there is no marked improvement in ventricular function following the injection/infusion of autologous mitochondria and the subject has a clinically indicated procedure in the days following the initial delivery, a second injection/infusion will be completed. At this time the follow up schedule will be reset to Day 0.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric cardiology patients under the age of 18 on ECMO
* concerns for ischemic injury on the Cardiac Intensive Care Unit

Exclusion Criteria:

* Known mitochondria disorders

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety- Incidence of severe adverse events | 1 week
  Subjects will be SAE free for one week following injection

SECONDARY OUTCOMES:
Efficacy- Improvement in Outcome measures: increased ventricular function on echocardiogram, measured by ejection fraction | 1 week- 1 month
  Improvement in ventricular function
Efficacy- Improvement in Outcome measures: ability to be separated from ECMO support, measured in days since injection | 1 week- 1 month
  The ability to decannulate from ECMO support

CONTACTS AND LOCATIONS:
Overall Officials: Sitaram M Emani, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided